CLINICAL TRIAL: NCT00431548
Title: Retinal Oxygen Reactivity in Patients Infected With Human Immunodeficiency Virus (HIV).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPHT-180198
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-02-06 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections; Retina; Ocular Physiology
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: 100% O2

SUMMARY:
Ocular lesions, including cotton wool spots and retinal hemorrhage, are a common feature of HIV infection and acquired immunodeficiency syndrome (AIDS). The aetiology of these apparently vasoocclusive phenomena in HIV related retinopathy is not well understood. Several hypotheses including infectious damage of the retinal vasculature and altered retinal hemodynamics have been postulated. The latter would be compatible with the theory that the retina of HIV patients is hypoxic. However, direct measurement of oxygen tension in the retina is not possible and indirect methods have to be employed. The study objective was to investigate the reactivity in retinal blood flow to 100% oxygen breathing in patients with HIV.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Patients with HIV)

* Aged between 19 and 70 years, male and female
* HIV positive patients without HIV-related retinopathy with a CD4+ cell count  500 cells/mm3 stage A2, A3, B2, B3, C2 and C3.
* Best corrected visual acuity >= 0.8
* Ametropy < 6 dpt

Group 2 (Healthy control subjects)

* Aged between 19 and 70 years
* Age and sex matched to the subjects in the HIV group (group matched)
* Matched with regard to the smoking habits in the HIV group
* Best corrected visual acuity >= 0.8
* Ametropy < 6 dpt

Exclusion Criteria:

* Evidence of any other eye disease
* Diabetes mellitus
* Systemic hypertension (defined as SBP > 150 mmHg or DBP > 90 mmHg)
* Abuse of illegal drugs

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30

PRIMARY OUTCOMES:
Reactivity in retinal blood flow during 100% O2 breathing expressed as percent change

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Eichler, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria